CLINICAL TRIAL: NCT07317804
Title: Comparison of Transcatheter Aortic Valve Replacement Using Echo Only With Echo Combined With X Ray for Patients With Aortic Stenosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Xiaopeng Hu, Principal Investigator, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-2761
Record Dates: First submitted 2025-12-11; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Aortic Stenosis; TAVI; TAVI(Transcatheter Aortic Valve Implantation)
Keywords: Ultrasound-guided; Percutaneous Intervention; TAVI(Transcatheter Aortic Valve Implantation); TAVI; Aortic Stenosis; PAN Procedure; non fluoroscopic
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echocardiography-guided group (Experimental): Patients randomized to the echocardiography-guided group will undergo a TAVI procedure under solely echo guidance.
  Interventions: Device: Echocardiographic guidance
- Fluoroscopy-guided intervention (Active Comparator): Patients randomized to the fluoroscopy-guided group will undergo a TAVI procedure under the combined guidance of X-ray and echo.
  Interventions: Device: Fluoroscopic guidance

INTERVENTIONS:
Device: Echocardiographic guidance — After detailed evaluation, patients randomized in this group will undergo TAVI procedure under guidance of fully echocardiography but any fluoroscopy in the entire process.
  Arms: Echocardiography-guided group
Device: Fluoroscopic guidance — After detailed evaluation, patients randomized in this group will undergo TAVI procedure under combined guidance of echocardiography and fluoroscopy in the entire process.
  Arms: Fluoroscopy-guided intervention

SUMMARY:
Aortic stenosis (AS) is a common valvular heart disease whose prevalence increases markedly with age-approximately 2-4% in individuals aged 65 years and older, and up to 3.4% for severe AS in those over 75. Degenerative calcific AS predominates in high-income countries, whereas rheumatic disease remains a major cause in low-income regions. With global population aging, the disease burden of AS continues to rise.

Transcatheter aortic valve replacement (TAVR/TAVI), owing to its minimally invasive nature, has become an important treatment option for severe AS and selected aortic regurgitation patients, expanding from high-surgical-risk populations to those at intermediate and low risk. In recent years, the number of TAVR procedures in many regions has surpassed or approached that of surgical aortic valve replacement, and major clinical guidelines have elevated TAVR to a recommended standard therapy.

Conventional TAVR relies on combined fluoroscopic and echocardiographic guidance. However, perioperative complications remain frequent in elderly and high-risk patients, particularly acute kidney injury (AKI), which significantly increases short- and long-term mortality. Contrast exposure during the procedure is a major contributor to AKI; thus, clinical practice increasingly favors strategies that minimize contrast use, such as low-dose and low-kV imaging. Elevated contrast concentration in the renal tubules increases viscosity, prolongs renal exposure, and can lead to tubular injury and renal dysfunction. Continuous radiation exposure during vascular access, device positioning, valve deployment, and post-release assessment also poses safety concerns for both patients and medical staff.

Echocardiography-only guidance for TAVR has therefore emerged as an attractive alternative, with the potential to replace fluoroscopy and contrast for anatomical visualization and device positioning, thereby reducing radiation exposure and contrast-related kidney injury. However, no prospective randomized study has directly compared echocardiography-only guidance with conventional fluoroscopy-plus-echocardiography guidance, and current evidence remains preliminary.

To address this gap, a randomized controlled trial was designed to evaluate whether echocardiography-only guidance is non-inferior to combined fluoroscopic and echocardiographic guidance in terms of device success, while also assessing the safety, efficacy, and clinical feasibility of both approaches.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 75 years or older with obvious clinical symptoms or a left ventricular ejection fraction less than 50% due to severe aortic valve stenosis (aortic valve orifice area < 1.0 cm² or peak velocity ≥ 4.0 m/s or mean transvalvular pressure ≥ 40 mmHg); or patients with obvious clinical symptoms of low blood flow and low pressure difference aortic valve stenosis (effective aortic valve orifice area < 1.0 cm², mean transvalvular pressure difference < 40 mmHg, left ventricular ejection fraction < 50%, stroke volume index < 35 ml/m², and diagnosed as true severe aortic valve stenosis by dobutamine stress test);
* 2. Patients aged 75 years > age ≥ 65 years with severe aortic stenosis who have surgical contraindications or high risks, or have other risk factors such as post-chest radiotherapy, liver failure, diffuse severe aortic calcification, extreme weakness, etc., or patients refuse to undergo routine open-chest surgery;
* 3. The patient's anatomical structure is suitable for TAVR and can tolerate transesophageal ultrasound;
* 4. The patient has signed the informed consent form and is willing to participate in this study.

Exclusion Criteria:

* 1. Imaging (ultrasound and/or CT and/or MRI) confirmed a lesion, thrombus or calculus in the left ventricle;
* 2. Severe obstruction of the left ventricular outflow tract;
* 3. Severe right ventricular dysfunction;
* 4. Acute myocardial infarction within 30 days before the surgery;
* 5. Active endocarditis history within 180 days before the surgery;
* 6. Inappropriate aortic root anatomy (such as combined aortic dissection, excessive aortic annulus, risk of coronary artery occlusion, etc.);
* 7. Severe calcification and distortion of the surgical approach;
* 8. Left ventricular ejection fraction less than 20%;
* 9. Other cardiac diseases that require concurrent treatment (such as severe mitral regurgitation, atrial fibrillation, etc.);
* 10. History of stroke or transient ischemic attack within 90 days before the surgery;
* 11. Liver cirrhosis or active liver disease;
* 12. Renal insufficiency (creatinine clearance rate < 30 mL/min) and/or undergoing renal replacement therapy;
* 13. Unable to tolerate anticoagulation therapy during or after the surgery;
* 14. Participating in other drug or device research;
* 15. Any emergency or surgical operation within 30 days before the surgery;
* 16. Other severe comorbidities, even if the valve stenosis is corrected, the expected life expectancy is less than 1 year;
* 17. Other conditions deemed unsuitable for TAVR surgery by the cardiac team.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The study adopted the definition of device success from the VARC-3 (Valve Academic Research Consortium - 3) and used the device success rate as the primary outcome measure. | at the time of the participants' discharge up to 15 days after the procedure
  Device success (at discharge) required the fulfillment of all of the following conditions:
  1. Technical success;
  2. No death;
  3. No additional surgery or intervention was required due to device-related, important vascular/pathway-related complications or cardiac structural complications related to the device (excluding permanent pacemakers);
  4. The valve achieved the expected performance (average transvalvular pressure difference < 20 mmHg, peak velocity < 3 m/s, Doppler velocity index ≥ 0.25, and no more than moderate-grade valve intra-aneurysmal reflux or paravalvular leakage).

SECONDARY OUTCOMES:
technique success | evaluated at the time of leaving the operating room
  technique success, according to the definition of technical success in the VARC-3, must meet all of the following conditions:
  1. No death;
  2. Successful establishment of vascular access, implantation of the valve, and withdrawal from the delivery system;
  3. Correct placement of a single artificial heart valve in the appropriate anatomical position;
  4. No surgical or interventional procedures due to complications from instruments, major blood vessels or access routes, or cardiac structures.
device success | at 30 days after the operation
  The 30-day device success rate was evaluated according to the definition of VARC-3 for device success. This metric must meet all of the following conditions:
  1. Technical success;
  2. No death;
  3. No surgical or interventional procedures due to complications from the device, main blood vessels or access, or cardiac structures;
  4. The valve achieves the expected performance (average transvalvular pressure gradient < 20 mmHg, peak velocity < 3 m/s, Doppler velocity index ≥ 0.25, and no more than moderate valve insufficiency or paravalvular leakage).
The all-cause mortality rate | at 30 days after the operation
  The all-cause mortality rate at 30 days after the operation
Cardiovascular mortality | at 30 days after the operation
  Cardiovascular mortality rate at 30 days after surgery
stroke | at 30 days after the operation
  The incidence of stroke 30 days after the operation
vascular complications | at 30 days after the operation
  The incidence of vascular complications 30 days after the operation
bleeding (including VARC-3 grade severe bleeding, life-threatening bleeding, and fatal bleeding) | at 30 days after the operation
  The incidence of postoperative bleeding (including VARC-3 grade severe bleeding, life-threatening bleeding, and fatal bleeding) at 30 days after surgery
acute kidney injury | at 30 days after the operation
  The incidence of acute kidney injury 30 days after the operation
The permanent pacemaker implantation(due to new conduction abnormalities or the aggravation of existing conduction abnormalities) | at 30 days after the operation
  The permanent pacemaker implantation rate 30 days after the surgery (due to new conduction abnormalities or the aggravation of existing conduction abnormalities)
coronary artery blockages that require intervention | at 30 days after the operation
  The incidence of coronary artery blockages that require intervention 30 days after the surgery
valve stenosis or regurgitation (perivalvular and central) | at 30 days after the operation
  At 30 days after the operation, echocardiography was used to assess the incidence of valve stenosis or regurgitation (perivalvular and central)
The re-hospitalization rate due to aortic valve stenosis or surgical complications within | at 30 days after the operation
  The re-hospitalization rate due to aortic valve stenosis or surgical complications within 30 days after the operation
new-onset atrial fibrillation | at 30 days after the operation
  The incidence of new-onset atrial fibrillation 30 days after the operation
structural valve regurgitation of the bioprosthetic aortic valve (as defined by VARC-3) | at 30 days after surgery
  The incidence of structural valve regurgitation of the bioprosthetic aortic valve (as defined by VARC-3) 30 days after surgery
time of operation | at discharge up to 15 days after procedure
  time of operation
Total hospital stay for TAVR surgery | at discharge up to 15 days after procedure
  Total hospital stay for TAVR surgery
fluoroscopy time | at discharge up to 15 days after procedure
  fluoroscopy time
Radiation dose | at discharge up to 15 days after procedure
  Radiation dose
Dose of contrast agent | at discharge up to 15 days after procedure
  Dose of contrast agent
hospital cost | at discharge up to 15 days after procedure
  Costs: Expenses related to the consumption of medical resources, such as costs of medical equipment and personnel; costs for hospitalization of research participants

CONTACTS AND LOCATIONS:
Overall Officials: Xiaopeng Hu, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing; Xiangbin Pan, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No